CLINICAL TRIAL: NCT02085161
Title: An Exploratory, 12 Week, Randomised, Partially Double-blinded, Placebo-controlled Parallel Group Trial to Explore the Effects of Once Daily Treatments of Orally Inhaled Tiotropium + Olodaterol Fixed Dose Combination or Tiotropium (Both Delivered by Respimat® Inhaler), Supervised Exercise Training and Behavior Modification on Exercise Capacity and Physical Activity in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: To Evaluate the Effect of Inhaled Medication Together With Exercise and Activity Training on Exercise Capacity and Daily Activities in Patients With Chronic Lung Disease With Obstruction of Airways
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1237.16; 2013-002671-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-07; First posted 2014-03-12 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — olodaterol; tiotropium-olodaterol; Tiotropium Bromide

ARMS (4):
- placebo (Placebo Comparator): patient will receive placebo once daily, 2 puffs in the morning
  Interventions: Drug: placebo to tiotropium + olodaterol
- tiotropium + olodaterol high dose with BM (Experimental): patient will receive tiotropium 5 mcg + olodaterol 5 mcg in fixed dose combination once daily, 2 puffs in the morning
  Interventions: Drug: tiotropium +olodaterol
- tiotropium (Active Comparator): patient will receive tiotropium 5 mcg once daily, 2 puffs in the morning
  Interventions: Drug: tiotropium
- tiotropium + olodaterol with exercise training and BM (Experimental): patient will receive tiotropium 5 mcg + olodaterol 5 mcg in fixed dose combination once daily, 2 puffs in the morning
  Interventions: Drug: tiotropium+olodaterol

INTERVENTIONS:
Drug: placebo to tiotropium + olodaterol — comparator
  Arms: placebo
Drug: tiotropium+olodaterol — tiotropium 5 mcg once daily
  Arms: tiotropium + olodaterol with exercise training and BM
Drug: tiotropium +olodaterol — olodaterol 5 mcg once daily fixed dose combination
  Arms: tiotropium + olodaterol high dose with BM
Drug: tiotropium — tiotropium 5 mcg once daily fixed dose combination
  Arms: tiotropium

SUMMARY:
The primary objectives of the study are to explore the effect of treatment with orally inhaled tiotropium + olodaterol fixed dose combination with and without exercise training, and tiotropium comparing to placebo, on top of behavioural modification in improving exercise capacity in patients with COPD

ELIGIBILITY:
Inclusion criteria:

* All patients must sign an informed consent consistent with International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) - Good Clinical Practice (GCP) guidelines prior to participation in the trial, which includes medication washout and restrictions.
* All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria: Patients must have relatively stable airway obstruction with a post-bronchodilator forced expiratory volume in one second >=30% and <80% of predicted normal; Global Initiative for Chronic Obstructive Lung Disease grade II - III, and a post-bronchodilator Tiffeneau index <70% at Visit 1.
* Male or female patients, aged >=40 years and <=75 years.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded.

Exclusion criteria:

* Patients with a significant disease other than chronic obstructive pulmonary disease.
* Patients with clinically relevant abnormal baseline haematology, blood chemistry, or urinalysis.
* Patients with a history of asthma.
* A diagnosis of thyrotoxicosis.
* A diagnosis of paroxysmal tachycardia (>100 beats per minute).
* A history of myocardial infarction within 1 year of screening visit.
* Unstable or life-threatening cardiac arrhythmia.
* Hospitalized for heart failure within the past year.
* Known active tuberculosis.
* A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years.
* A history of life-threatening pulmonary obstruction and patients with chronic respiratory failure.
* A history of cystic fibrosis.
* Clinically evident bronchiectasis.
* A history of significant alcohol or drug abuse.
* Any contraindications for exercise testing.
* Patients who have undergone thoracotomy with pulmonary resection.
* Patients being treated with any oral ß-adrenergics.
* Patients being treated with oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose) or at doses in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day.
* Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigators opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit or patients who are currently in a pulmonary rehabilitation program.
* Patients who have a limitation of exercise performance as a result of factors other than fatigue or exertional dyspnoea, such as arthritis in the leg, angina pectoris or claudication or morbid obesity.
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to screening visit.
* Patients with known hypersensitivity to ß-adrenergics drugs, anticholinergic drugs, benzalkonium chloride, disodium edentat, or any other component of the Respimat® inhalation solution delivery system.
* Pregnant or nursing women.
* Women of childbearing potential not using highly effective methods of birth control.
* Patients who have previously been randomized in this study or are currently participating in another study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (34):
- United States (3):
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - Boehringer Ingelheim Investigational Site, Torrance, California
  - Boehringer Ingelheim Investigational Site, Hartford, Connecticut
- Australia (2):
  - Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - Boehringer Ingelheim Investigational Site, Glen Osmond, South Australia
- Boehringer Ingelheim Investigational Site, Salzburg, Austria
- Belgium (3):
  - Boehringer Ingelheim Investigational Site, Genk
  - Boehringer Ingelheim Investigational Site, Hasselt
  - Boehringer Ingelheim Investigational Site, Leuven
- Canada (3):
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Boehringer Ingelheim Investigational Site, Ste-Foy, Quebec
  - Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Denmark (3):
  - Boehringer Ingelheim Investigational Site, Kolding
  - Boehringer Ingelheim Investigational Site, København NV
  - Boehringer Ingelheim Investigational Site, Odense
- Germany (9):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Bochum
  - Boehringer Ingelheim Investigational Site, Frankfurt
  - Boehringer Ingelheim Investigational Site, Großhansdorf
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Leverkusen
  - Boehringer Ingelheim Investigational Site, Solingen
  - Boehringer Ingelheim Investigational Site, Teuchern
  - Boehringer Ingelheim Investigational Site, Tübingen
- Boehringer Ingelheim Investigational Site, Greenlane East Auckland NZ, New Zealand
- Poland (3):
  - Boehringer Ingelheim Investigational Site, Gdansk
  - Boehringer Ingelheim Investigational Site, Lodz
  - Boehringer Ingelheim Investigational Site, Starachowice
- Portugal (3):
  - Boehringer Ingelheim Investigational Site, Coimbra
  - Boehringer Ingelheim Investigational Site, Lisbon
  - Boehringer Ingelheim Investigational Site, Porto
- United Kingdom (3):
  - Boehringer Ingelheim Investigational Site, Leicester
  - Boehringer Ingelheim Investigational Site, Norwich
  - Boehringer Ingelheim Investigational Site, Sheffield

REFERENCES:
- [Derived] Troosters T, Bourbeau J, Maltais F, Leidy N, Erzen D, De Sousa D, Korducki L, Hamilton A. Enhancing exercise tolerance and physical activity in COPD with combined pharmacological and non-pharmacological interventions: PHYSACTO randomised, placebo-controlled study design. BMJ Open. 2016 Apr 13;6(4):e010106. doi: 10.1136/bmjopen-2015-010106. PMID 27075841
- [Derived] Bourbeau J, Lavoie KL, Sedeno M, De Sousa D, Erzen D, Hamilton A, Maltais F, Troosters T, Leidy N. Behaviour-change intervention in a multicentre, randomised, placebo-controlled COPD study: methodological considerations and implementation. BMJ Open. 2016 Apr 4;6(4):e010109. doi: 10.1136/bmjopen-2015-010109. PMID 27044576

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An exploratory, randomised, partially double-blinded, placebo-controlled, parallel group trial to explore the effects of tiotropium + olodaterol fixed dose combination (FDC) or tiotropium, supervised exercise training and behaviour modification on exercise capacity and physical activity in patients with Chronic Obstructive Pulmonary Disease (COPD)
Groups:
- Placebo With Behavioural Modification (BM): Placebo matching tiotropium + olodaterol FDC or tiotropium solution was delivered to the patients orally once daily via RESPIMAT inhaler, with BM for 12 weeks.
- Tiotropium (Tio) 5 Micro-grams (μg) With BM: Tiotropium 5 μg solution was delivered to the patients orally once daily via RESPIMAT inhaler, with BM for 12 weeks.
- Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM: Tiotropium 5 μg plus olodaterol 5 μg FDC solution was delivered to the patients orally once daily via RESPIMAT inhaler, with BM for 12 weeks.
- Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM: Tiotropium 5 μg plus olodaterol 5 μg FDC solution was delivered to the patients orally once daily via RESPIMAT inhaler, with BM for 12 weeks; ET was conducted for 8 weeks.
Period: Overall Study
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Started | 76 | 76 | 76 | 76
Completed | 64 | 66 | 71 | 66
Not Completed | 12 | 10 | 5 | 10
Not completed — Not Treated | 1 | 0 | 0 | 0
Not completed — Adverse Event | 8 | 5 | 4 | 5
Not completed — Protocol Violation | 0 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 4 | 0 | 3
Not completed — Other Reason | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set included all patients of the Randomised set (All patients who signed informed consent form and were also randomised, regardless whether the patient was treated with study medication or not.) who were dispensed study medication and were documented to have taken any dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM | Total
Number analyzed (Participants) | 75 | 76 | 76 | 76 | 303
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (6.6) | 65.1 (6.4) | 65.0 (6.9) | 64.7 (6.5) | 64.8 (6.6)
Gender [Count of Participants; unit: Participants]
  Female | 23 | 21 | 28 | 31 | 103
  Male | 52 | 55 | 48 | 45 | 200

OUTCOME MEASURES:

1. Primary Outcome: Endurance Time During Endurance Shuttle Walk Test (ESWT) to Symptom Limitation After 8 Weeks
Description: Endurance time during ESWT to symptom limitation at walking speed corresponding to 85% of predicted maximum oxygen consumption (VO2 peak) after 8 weeks of pharmacological treatment and non-pharmacological intervention. The numerical value of endurance time in seconds was transformed in log10 scale to correct for skewness and then an analysis of covariance (ANCOVA) was fitted to the log10-transformed data and the least square means (LSMean) and standard error (SE) were obtained. To present the results in a way easier for interpretation, the least square mean from the ANCOVA fitted to the log10-transformed data were transformed back taking 10 to the power of the least square estimate to obtain the geometric mean and the corresponding SE was transformed using delta method to get the corresponding SE of the geometric mean.
Time Frame: Week 8
Population: Full analysis set (FAS): This patient set included all patients in the Treated set (TS) who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint. Patients were assigned to the FAS after implementation of any data handling rules that set measurements to missing. Patients with available data were included.
Measure: Geometric Mean (Standard Error); unit: Second
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 65 | 67 | 72 | 70
Second | 244.07 (17.666) | 254.18 (18.099) | 315.32 (21.671) | 355.73 (24.787)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; This treatment comparison is the first one in the alpha-protected hierarchical testing chain; Test type: Superiority or Other; p = 0.0002, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; Mean and 95% confidence limits were transformed from log10 back to the original scale. SE was back transformed using the delta method; Treatment ratio = 1.458, 95% CI 2-sided [1.196 to 1.777], Standard Error of Mean 0.147 — Ratio of means calculated as back transformation of difference on log 10 scale between Tio+Olo (5/5 μg) FDC with exercise training (ET) and BM minus Placebo with behavioural modification (BM)
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; This treatment comparison is the second one in the alpha-protected hierarchical testing chain; Test type: Superiority or Other; p = 0.0109, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.292, 95% CI 2-sided [1.061 to 1.573], Standard Error of Mean 0.129 — Ratio of means calculated as back transformation of difference on log 10 scale between Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM minus Placebo with behavioural modification (BM)
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; This treatment comparison is the third one in the alpha-protected hierarchical testing chain. Since the p-value for this treatment comparison is >0.05, the hierarchical testing chain is broken and all of the following hypothesis tests in this hierarchical chain are considered as descriptive only; Test type: Superiority or Other; p = 0.6895, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.041, 95% CI 2-sided [0.853 to 1.272], Standard Error of Mean 0.106 — Ratio of means calculated as back transformation of difference on log 10 scale between Tiotropium (Tio) 5 micro-grams (μg) with BM minus Placebo with behavioural modification (BM)
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.2188, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.128, 95% CI 2-sided [0.931 to 1.368], Standard Error of Mean 0.110 — Ratio of means calculated as back transformation of difference on log 10 scale between Tio+Olo (5/5 μg) FDC with exercise training (ET) and BM minus Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0303, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.241, 95% CI 2-sided [1.021 to 1.507], Standard Error of Mean 0.123 — Ratio of means calculated as back transformation of difference on log 10 scale between Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM minus Tiotropium (Tio) 5 micro-grams (μg) with BM

2. Secondary Outcome: Average Daily Walking Time Measured by the Activity Monitor in the Week Prior to Week 12
Description: Average daily walking time measured by the activity monitor in the week prior to Week 12.
Time Frame: Week 12
Population: Full analysis set (FAS): This patient set included all patients in the TS who had baseline measurement and at least 1 post-baseline measurement for the primary endpoint. Patients were assigned to the FAS after implementation of any data handling rules that set measurements to missing. Patients with available data were included.
Measure: Least Squares Mean (Standard Error); unit: Second
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 55 | 57 | 60 | 57
Second | 4670.78 (211.798) | 4145.85 (207.351) | 4831.85 (202.261) | 4338.80 (207.252)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.2639, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -331.975, 95% CI 2-sided [-916.015 to 252.064], Standard Error of Mean 296.375 — The LSMean Difference is calculated as Tio+Olo (5/5 μg) FDC with exercise training (ET) and BM minus Placebo with behavioural modification (BM)
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.5837, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 161.072, 95% CI 2-sided [-417.314 to 739.459], Standard Error of Mean 293.506 — The LSMean Difference is calculated as Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM minus Placebo with behavioural modification (BM)
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p = 0.0783, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -524.926, 95% CI 2-sided [-1109.806 to 59.954], Standard Error of Mean 296.802 — The LSMean Difference is calculated as Tiotropium (Tio) 5 micro-grams (μg) with BM minus Placebo with behavioural modification (BM)
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.0900, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -493.048, 95% CI 2-sided [-1063.670 to 77.575], Standard Error of Mean 289.566 — The LSMean Difference is calculated as Tio+Olo (5/5 μg) FDC with exercise training (ET) and BM minus Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0186, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 685.998, 95% CI 2-sided [115.635 to 1256.362], Standard Error of Mean 289.435 — The LSMean Difference is calculated as Tiotropium + olodaterol (Olo) (5/5 μg) FDC with BM minus Tiotropium (Tio) 5 micro-grams (μg) with BM

3. Secondary Outcome: Average Daily Walking Intensity Measured by the Activity Monitor in the Week Prior to 12 Weeks of Treatment
Description: Average daily walking intensity measured by the activity monitor in the week prior to 12 weeks of treatment. The Movement Intensity (MI) is derived from the acceleration signals. Since seismic sensors measure gravitational acceleration (g) in static situations, the acceleration signal is expressed relative to g (1g = 9.81m/s2). To calculate movement intensity (MI) the gravitational acceleration in static situations was removed and the rotation vector of the three accelerometer signals was calculated. The MI gives an indication of the power of movements.
Time Frame: Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Multiple of 9.8*(meters / (second^2))
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 54 | 56 | 58 | 57
Multiple of 9.8*(meters / (second^2)) | 0.20 (0.003) | 0.20 (0.003) | 0.20 (0.003) | 0.20 (0.003)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.5186, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -0.002, 95% CI 2-sided [-0.010 to 0.005], Standard Error of Mean 0.004 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.6436, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.002, 95% CI 2-sided [-0.006 to 0.009], Standard Error of Mean 0.004 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p = 0.1081, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -0.006, 95% CI 2-sided [-0.014 to 0.001], Standard Error of Mean 0.004 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.2612, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -0.004, 95% CI 2-sided [-0.011 to 0.003], Standard Error of Mean 0.004 — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0361, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.008, 95% CI 2-sided [0.001 to 0.015], Standard Error of Mean 0.004 — [estimate comment as in outcome 2, analysis 5]

4. Secondary Outcome: Perceived Difficulties as Evaluated With Functional Performance Inventory-Short Form (FPI-SF) Total Score at Week 12
Description: Perceived difficulties as evaluated with FPI-SF. FPI-SF self-report questionnaire has 6 domains: Body care(5 items), Household maintenance(8 items), Physical exercise(5 items), Recreation(5 items), Spiritual activities(4 items) and Social interaction(5 items) with five possible answers on each item: Do with no difficulty - 3, Do with some difficulty - 2, Do with great difficulty - 1, don't do because of health reasons - 0, and don't do because choose not to - 0. Domain scores are expressed as mean values, with at least 6 non-missing items required for the household maintenance domain and at least 3 non-missing items for the other domains. Total score is the mean across the six domains. So total and domain scores range from 0 to 3, with higher scores indicating higher levels of functional activity within and across domains. Respondents engaged in many activities with no difficulty will score high on the FPI, while those who perform few activities with much difficulty will score low.
Time Frame: Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 64 | 65 | 71 | 67
Units on a scale | 2.191 (0.040) | 2.207 (0.040) | 2.335 (0.038) | 2.268 (0.039)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.1727, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.076, 95% CI 2-sided [-0.034 to 0.187], Standard Error of Mean 0.056 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0097, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.143, 95% CI 2-sided [0.035 to 0.252], Standard Error of Mean 0.055 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p = 0.7815, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.016, 95% CI 2-sided [-0.095 to 0.126], Standard Error of Mean 0.056 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.2183, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = -0.067, 95% CI 2-sided [-0.174 to 0.040], Standard Error of Mean 0.054 — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0203, ANCOVA — An ANCOVA model with categorical effects of treatment and baseline as covariate; LSMean Difference = 0.128, 95% CI 2-sided [0.020 to 0.236], Standard Error of Mean 0.055 — [estimate comment as in outcome 2, analysis 5]

5. Secondary Outcome: Endurance Time During Endurance Shuttle Walk Test (ESWT) to Symptom Limitation After 12 Weeks
Description: Endurance time during ESWT to symptom limitation at walking speed corresponding to 85% of maximum oxygen consumption (VO2 peak) after 12 weeks of pharmacological treatment and non-pharmacological intervention. The numerical value of endurance time in seconds was transformed in log10 scale to correct for skewness and then the ANCOVA was fitted to the log10-transformed data and the least square means and SE were obtained. To present the results in a way easier for interpretation, the least square mean from the ANCOVA fitted to the log10-transformed data were transformed back taking 10 to the power of the least square estimate to obtain the geometric mean and the corresponding SE was transformed using delta method to get the corresponding SE of the geometric mean.
Time Frame: Week 12
Population: as for outcome 2
Measure: Geometric Mean (Standard Error); unit: Second
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 62 | 64 | 71 | 66
Second | 243.30 (18.680) | 255.67 (19.292) | 302.61 (21.691) | 324.21 (24.095)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.0077, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.333, 95% CI 2-sided [1.080 to 1.645], Standard Error of Mean 0.142 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0390, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.244, 95% CI 2-sided [1.011 to 1.530], Standard Error of Mean 0.131 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p = 0.6452, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.051, 95% CI 2-sided [0.850 to 1.299], Standard Error of Mean 0.113 — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.5048, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.071, 95% CI 2-sided [0.874 to 1.313], Standard Error of Mean 0.111 — [estimate comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.1066, ANCOVA — ANCOVA model with categorical effect of treatment and baseline as covariate; [statistical method as in outcome 1, analysis 1]; Treatment ratio = 1.184, 95% CI 2-sided [0.964 to 1.453], Standard Error of Mean 0.123 — [estimate comment as in outcome 1, analysis 5]

6. Secondary Outcome: One Hour, Post-dose Forced Expiratory Volume in One Second (FEV1) After 8 Weeks of Treatment
Description: One hour, Post-dose Forced Expiratory Volume in One Second (FEV1) after 8 weeks of treatment.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 65 | 67 | 72 | 70
Liter | 1.375 (0.027) | 1.550 (0.027) | 1.731 (0.026) | 1.705 (0.026)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — Mixed effect Model Repeat Measurement (MMRM) including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; Compound symmetry covariance structure for within-patient variation and Kenward-Roger approximation of denominator degrees of freedom; LSMean Difference = 0.329, 95% CI 2-sided [0.255 to 0.403], Standard Error of Mean 0.038 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — MMRM model including fixed effects of treatment, planned test day, treatment by test day interaction, baseline, and baseline by test day interaction; patient as a random effect; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.356, 95% CI 2-sided [0.282 to 0.429], Standard Error of Mean 0.037 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.174, 95% CI 2-sided [0.099 to 0.249], Standard Error of Mean 0.038 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.4677, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = -0.027, 95% CI 2-sided [-0.099 to 0.045], Standard Error of Mean 0.037 — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.182, 95% CI 2-sided [0.109 to 0.255], Standard Error of Mean 0.037 — [estimate comment as in outcome 2, analysis 5]

7. Secondary Outcome: One Hour, Post-dose Forced Vital Capacity (FVC) After 8 Weeks of Treatment
Description: One hour, Post-dose Forced Vital Capacity (FVC) after 8 weeks of treatment.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 65 | 67 | 72 | 70
Liter | 2.974 (0.047) | 3.259 (0.046) | 3.504 (0.044) | 3.452 (0.045)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.478, 95% CI 2-sided [0.350 to 0.606], Standard Error of Mean 0.065 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.530, 95% CI 2-sided [0.403 to 0.657], Standard Error of Mean 0.064 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.286, 95% CI 2-sided [0.157 to 0.415], Standard Error of Mean 0.066 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.4107, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = -0.052, 95% CI 2-sided [-0.176 to 0.072], Standard Error of Mean 0.063 — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0002, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.244, 95% CI 2-sided [0.119 to 0.370], Standard Error of Mean 0.064 — [estimate comment as in outcome 2, analysis 5]

8. Secondary Outcome: Resting Inspiratory Capacity (IC) Measured at 1.5 Hours Post Dose After 8 Weeks of Treatment
Description: Resting inspiratory capacity (IC) measured at 1.5 hours post dose after 8 weeks of treatment.
Time Frame: Week 8
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM
Number analyzed (Participants) | 64 | 66 | 72 | 68
Liter | 2.452 (0.051) | 2.627 (0.050) | 2.755 (0.048) | 2.771 (0.049)
Statistical Analysis 1: Comparison: Placebo With Behavioural Modification (BM) vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 1]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.318, 95% CI 2-sided [0.179 to 0.457], Standard Error of Mean 0.071 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.302, 95% CI 2-sided [0.165 to 0.439], Standard Error of Mean 0.070 — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Placebo With Behavioural Modification (BM) vs Tiotropium (Tio) 5 Micro-grams (μg) With BM; Test type: Superiority or Other; p = 0.0145, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.174, 95% CI 2-sided [0.035 to 0.314], Standard Error of Mean 0.071 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 4: Comparison: Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM vs Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM; Test type: Superiority or Other; p = 0.8150, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.016, 95% CI 2-sided [-0.118 to 0.151], Standard Error of Mean 0.068 — [estimate comment as in outcome 2, analysis 4]
Statistical Analysis 5: Comparison: Tiotropium (Tio) 5 Micro-grams (μg) With BM vs Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM; Test type: Superiority or Other; p = 0.0642, Mixed Models Analysis — [p-value comment as in outcome 6, analysis 2]; [statistical method as in outcome 6, analysis 1]; LSMean Difference = 0.128, 95% CI 2-sided [-0.008 to 0.263], Standard Error of Mean 0.069 — [estimate comment as in outcome 2, analysis 5]

ADVERSE EVENTS:
Time Frame: From first dose of study medication up to a period of 21 days after the last dose of study medication were assigned to the treatment period, up to 134 days.
Description: All adverse events, serious and non-serious, occurring during the course of the clinical trial (i.e. from signing the informed consent onwards through the observational phase) were to be collected, documented and reported to the sponsor by the investigator on the appropriate electronic case report form / serious adverse event reporting forms.
Groups:
- Total: Total
Arm/Group | Placebo With Behavioural Modification (BM) | Tiotropium (Tio) 5 Micro-grams (μg) With BM | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM | Total
Serious Adverse Events (participants affected / at risk) | 4/75 | 11/76 | 3/76 | 8/76 | 26/303
Other Adverse Events (participants affected / at risk) | 22/75 | 19/76 | 16/76 | 19/76 | 76/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Behavioural Modification (BM) (N=75) | Tiotropium (Tio) 5 Micro-grams (μg) With BM (N=76) | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM (N=76) | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM (N=76) | Total (N=303)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Malignant genitourinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Non-Hodgkin's lymphoma unspecified histology indolent stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo With Behavioural Modification (BM) (N=75) | Tiotropium (Tio) 5 Micro-grams (μg) With BM (N=76) | Tiotropium + Olodaterol (Olo) (5/5 μg) FDC With BM (N=76) | Tio+Olo (5/5 μg) FDC With Exercise Training (ET) and BM (N=76) | Total (N=303)
Nasopharyngitis (Infections and infestations) | 8 | 9 | 4 | 10 | 31
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1 | 8
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 | 10 | 12 | 13 | 51
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2 | 2 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.